CLINICAL TRIAL: NCT03625453
Title: A Randomized, Placebo-Controlled Study of ABX-1431 in Adult Patients With Tourette Syndrome or Chronic Motor Tic Disorder
Brief Title: Study of ABX-1431 in Adult Patients With Tourette Syndrome or Chronic Motor Tic Disorder
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Abide Therapeutics (Industry)
Collaborators: FGK Clinical Research GmbH (Industry); BASi (Bioanalytical Systems, Inc.) (Industry); CogState Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ABX-1431 PN018; 2018-000100-41 (EudraCT Number)
Record Dates: First submitted 2018-08-08; First posted 2018-08-10 (Actual); Last update posted 2020-04-08 (Actual); Status verified 2020-04

CONDITIONS: Tourette Syndrome; Motor Tic Disorder
Keywords: Tourette Syndrome; Chronic Motor Tic Disorder
MeSH Terms: conditions — Tourette Syndrome; Tic Disorders | interventions — ABX-1431

STUDY DESIGN:
Intervention Model Description: Randomized, placebo-controlled
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ABX-1431 (Experimental): Oral use of hard capsule (10 milligrams), maximum dose per day: 40 milligrams
  Interventions: Drug: ABX-1431
- Placebo (Placebo Comparator): Oral use of hard capsule
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ABX-1431 — Part 1: 8 weeks with daily administration; Patients who choose to enter Part 2: additional 4 weeks with daily administration
  Arms: ABX-1431
Drug: Placebo — Part 1: 8 weeks with daily administration
  Arms: Placebo

SUMMARY:
Two-part study consisting of a double-blind, randomized, placebo-controlled, study at two target dose levels (Part 1) and an open-label, non-randomized study (Part 2) to determine the efficacy of ABX-1431 in treating adult patients with Tourette syndrome or Chronic Motor Tic Disorder as measured by the change from baseline in Total Tic Score of the Yale Global Tic Severity Scale (YGTSS-TTS) compared with placebo.

DETAILED DESCRIPTION:
ABX-1431 is a potent and selective, orally available, irreversible inhibitor of monoacylglycerol lipase, a metabolic enzyme that regulates the activity of the endogenous cannabinoid (endocannabinoid) system. It is being developed as a potential first-in-class compound for the treatment of Tourette Syndrome.

This study will assess the safety, tolerability, and effect on tics ABX-1431 in adults with Tourette Syndrome or chronic motor tic disorder in an 8-week study. It is a two-part study. Part 1 is a double-blind, randomized, placebo-controlled study of ABX-1431 at two target dose levels. Part 2 is an optional, open-label, non-randomized study of ABX-1431.

Patients will participate in the main study (Part 1) for approximately 10 to 14 weeks (up to 30-day screening period; 56-day treatment period; 14-day follow-up period). For patients who choose to participate in Part 2, there is a period of up to 4 weeks between the last study visit in Part 1 and first study visit in Part 2. Patients who choose to enter Part 2 will be treated with open-label ABX-1431 for an additional 6 weeks (28-day treatment period; 14-day follow-up period).

ELIGIBILITY:
Inclusion Criteria:

1. Patient is a male or female ≥ 18 to 64 years of age at the Screening Visit.
2. Patient has a diagnosis of Tourette Syndrome or Chronic Motor Tic Disorder as defined by the Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5) criteria.
3. Patient's YGTSS-TTS results must be ≥ 22 (range 0-50) at the Baseline/Randomization Visit.
4. At the Baseline/Randomization Visit patients must be taking a stable drug regimen for tics and comorbidities for 30 days and must be expected to remain on a stable drug regimen during this study. Patients receiving no medication for TS may participate. Patients who have recently discontinued medication for tics must have discontinued them for at least 30 days. For neuroleptic drugs (e.g., risperidone, aripiprazole), the minimum discontinuation period is 30 days prior to the Baseline/Randomization Visit. For injectable depot neuroleptic drugs the minimum discontinuation period is one dosage cycle plus 14 days. (See Inclusion 'f' for discontinuation period of cannabinoid medication in patients using these products for tics.)
5. Patient is legally competent, has been informed of the nature and scope of relevance for the study, voluntarily agrees to participation, agrees to the study restrictions, and has signed the informed consent form (ICF) approved by the Ethics Review Committee (ERC).
6. Patients using cannabinoid medications for their tics must discontinue their use at least 14 days prior to the Baseline/Randomization Visit. The investigator and patient must be confident that these patients will not require these medications for the duration of the study until 14 days after the last dose of study medication. Examples of cannabinoids include cannabis in any form, nabilone or Δ9-tetrahydrocannabinol (THC)-containing medications such as nabiximols (Sativex®) or dronabinol. The use of recreational cannabinoids during this study is not permitted.
7. Female patients of child-bearing potential must have a negative pregnancy test [serum or urine human chorionic gonadotropin (hCG)] at the Screening Visit and other indicated visits. They must practice a highly effective, reliable, and medically approved contraceptive regimen during the study (e.g., theoretical failure rate less than 1% per year as described in the 2014 Heads of Medicines Agencies: Clinical Trials Facilitation Group report on contraception in clinical trials, which include oral or parenteral or implanted hormonal contraception, vaginal ring releasing hormonal contraception (e.g., Nuvaring, intrauterine device, or intrauterine system). Post-menopausal women may enter this study. Post-menopausal women are defined as those without menses in the past 12 months, and with a serum follicle stimulating hormone (FSH) in the post-menopausal range. Women who are surgically sterile may enter this study with written documentation of the surgical procedure.
8. Male patients must be willing to use a condom with sexual partners during this study until 14 days after the last dose of study medication. Male patients must be willing to abstain from sperm donation for 3 months after the completion of this study.

Exclusion Criteria:

1. Patient is taking strong inducers or inhibitors of cytochrome P450 (CYP)3A4/5 or CYP2C9. Examples of strong CYP3A4/5 inducers include carbamazepine, efavirenz, nevirapine, barbiturates, pioglitazone, modafinil, enzalutamide, oxcarbazepine, rifampicin, St. John's Wort (Hypericum perforatum), and phenytoin. Examples of potent CYP3A4/5 inhibitors include atazanavir, boceprevir, clarithromycin, grapefruit juice, indinavir, itraconazole, ketoconazole, nefazodone, suboxone, nelfinavir, posaconazole, ritonavir, saquinavir, telithromycin, and voriconazole. Examples of CYP2C9 strong inducers/inhibitors include carbamazepine, enzalutamide, fluconazole, valproic acid, phenobarbital, nevirapine, rifampicin, and St. John's Wort.
2. Patient has evidence of alcohol abuse or dependence, as defined by the DSM-5 criteria, with two or more of the 11 criteria at the Screening Visit or within 1 year before the Screening Visit.
3. Patient has evidence of drug or chemical abuse (except nicotine), as defined by the DSM-5 criteria, at the Screening Visit or within 1 year before the Screening Visit. Patient has evidence of marijuana or cannabis dependency or has been treated for cannabis dependency, as defined by DSM-5 criteria, at the Screening Visit or within 1 year before the Screening Visit. (Patients who are prescribed stimulants should not be assessed for Stimulant Use Disorder. Patients who use cannabinoid-based medicine (e.g., cannabis in any form, nabilone, or THC-containing medications) for treatment of Tourette Syndrome with the investigator's knowledge should not be assessed for Cannabis Use Disorder, but these patients must comply with abstinence requirements for this study (See Inclusion 'f')). Patients who have a positive urine drug screen at the Screening Visit for drugs other than those allowed, as indicated in this criterion, are excluded.
4. Patient is unwilling to comply with study restrictions including abstinence from cannabis and alcohol from the Baseline/Randomization Visit until the follow-up telephone call 14 days after the last dose of study medication.
5. Patients receiving ongoing psychological therapy for tics such as Habit Reversal Training or Comprehensive Behavioral Intervention for Tics are excluded. Patients who have completed behavioral therapy for tics at least 30 days before the Baseline/Randomization Visit may participate.
6. Patient is a lactating or pregnant female, or a female who intends to become pregnant within 90 days following the last dose of study medication.
7. Patient has one or more of the following laboratory results at the Screening Visit:

   * Aspartate transaminase (AST) > 3 x upper limit of normal (ULN)
   * Alanine transaminase (ALT) > 3 x ULN
   * Total bilirubin > 2 x ULN (unless due to Gilbert's syndrome)
8. Patient has an estimated creatinine clearance less than 60 mL/minute at the Screening Visit. Creatinine clearance (Clcr) is estimated by the Cockcroft-Gault (C-G) equation from a spot serum creatinine (mg/dL) determination using the following formula:

   CLcr (mL/min) = [140 - age (years)] × weight (kg) / 72 × serum creatinine (mg/dL)] × [0.85 for female patients]
9. Patient has a serum albumin level below the laboratory normal range at the Screening Visit, and the physician cannot rule out hepatic insufficiency based on consideration of clinical symptoms, clinical signs, and other laboratory tests. (The physician may decide that a low value of a serum albumin is clinically insignificant or the test may be repeated.)
10. Patient has symptomatic chronic Hepatitis B and/or Hepatitis C Virus infection. Asymptomatic seropositive individuals without clinical or clinical laboratory manifestations of hepatitis may be enrolled.
11. Patient has a clinically significant abnormality on the ECG at the Screening Visit.
12. Patients with a history of cancer will be excluded, with two exceptions: Patients with a history of squamous or basal cell carcinoma of the skin treated with documented success of curative therapy > 3 months may be enrolled. Patients with cancer and in remission with no treatment for at least 2 years prior to the Screening Visit may be enrolled.
13. Patient has Tourette Syndrome or Chronic Motor Tic Disorder and also has mental retardation, autism spectrum disorder (ASD), dystonia, or post-traumatic stress disorder (PTSD). Mental retardation may be defined by medical history. (If the patient's available medical history is unclear, the investigator may use any validated screening test such as the Wechsler Abbreviated Scale of Intelligence (WASI-II); an intelligence quotient < 80 (well below average) is an exclusion). ASD and PTSD may be determined by medical history. (If the patient's available medical history is unclear, the investigator may use the diagnostic criteria for ASD and PTSD, as defined by the DSM-5.)
14. Patient has confounding medical conditions such as active infection, primary or acquired immunodeficiency (HIV testing is not mandated), uncontrolled diabetes (i.e., known Type 1 or 2 diabetes with most recent HbA1c level > 9.0% or has not had an HbA1c measurement within past 12 months), clinically significant cardiac disease (i.e., significant cardiac conduction abnormalities, uncontrolled hypertension, myocardial infarction, cardiac arrhythmia or unstable angina < 6 months to enrollment, New York Heart Association (NYHA) Grade II or greater congestive heart failure, serious cardiac arrhythmia requiring medication, Grade II or greater peripheral vascular disease, and history of cerebrovascular accident within 6 months), clinically significant renal disease (e.g., acute kidney injury (e.g., hematuria, oligouria, or an acute rise in serum creatinine of ≥ 0.5 mg / dL (≥ 44 umol/L)) or chronic kidney disease defined by estimated glomerular filtration rate < 60 ml / min or oligouria), or any suspected hepatic insufficiency. (See Exclusions 'g' 'h' and 'i' for laboratory test exclusion limits.) Physicians should rely on the medical history, physical examination, and protocol specified laboratory tests to exclude individuals with these conditions.
15. Patient has a diagnosis of any psychiatric comorbidity such obsessive compulsive disorder, attention deficit hyperactivity disorder, anxiety disorder, and/or depression and has undergone a change in therapy in the 30 days before the Baseline/Randomization Visit or is in need of a change in treatment. Patients with stable obsessive compulsive disorder or attention deficit hyperactivity disorder or depression requiring no alteration in therapy may be enrolled. Patients with a past history of psychosis or schizophrenia at any time are excluded.
16. Patient has a history of suicidal ideation with intent to act or a plan to act, or a suicide attempt in the last 3 years preceding the Baseline/Randomization Visit.
17. Patient has participated in an investigational study for medications with the last visit within 1 month for a non-biologic agent and 90 days for a biologic agent of the Baseline/Randomization Visit. The total volume of blood donated in the past 56 days may not exceed 450 mL.
18. Patient is an employee of the investigative site or sponsor or a close relative of an employee of the investigative site.
19. Patient has intolerance or hypersensitivity to the investigational medicinal product, ABX-1431 or the excipients. The excipients used in the capsule formulation are microcrystalline cellulose, croscarmellose sodium, magnesium stearate (vegetable origin), and gelatin capsule shells. The capsule shells are comprised of gelatin, red iron oxide, and titanium dioxide.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2018-10-15 (Actual); Primary Completion 2020-01-20 (Actual); Study Completion 2020-01-20 (Actual)

PRIMARY OUTCOMES:
Change from baseline in Total Tic Score of the Yale Global Tic Severity Scale (YGTSS-TTS) compared with placebo | Day 56 (40 mg ABX-1431 per day) and Day 28 (20 mg ABX-1431 per day)
  The Yale Global Tourette Severity Scale (YGTSS) is a clinician-completed rating scale to capture TS symptom severity. The number, frequency, intensity, complexity, and interference of both motor and vocal tics are rated on an ordinal scale between 0 and 5, with higher scores indicating greater severity. Motor and vocal tics subscales are reported (0 - 25) and then summed for a total tic score (TTS) (0 - 50). The TTS has been used as the registration endpoint for pharmacological therapies. The YGTSS has an Impairment subscale (0 - 50) which is then added for a total global score of 0 - 100.

SECONDARY OUTCOMES:
Adult Tic Questionnaire (ATQ) | Part 1: days 0, 14, 28, 42, 56; Part 2: days 0, 14, 28
  The Adult Tic Questionnaire (ATQ) is a tic self-rating scale. The ATQ records the occurrence, frequency and intensity for any of 27 endorsed common motor and vocal tics. The occurrence is being indicated as 1 for a present tic or 0 if no tic has been experienced. Frequency is measured on a scale from 1 (weekly frequency or less) to 4 (constant tics, almost all the time during the day). Intensity is being rated on a scale of 1 - 4 with 1 representing mild tics and 4 strong tics. The ATQ will principally be analyzed by summing the product of the intensity (1-4) and frequency (1-4) to determine the severity (2-8) across all endorsed tics. For clarity, the number of each endorsed tic and the total of intensity and frequency across all tics may be separately analyzed by mixed-model repeated-measures. The clinical relevance of changes in the ATQ may also be presented by the change in the average intensity and frequency score.
Premonitory Urge for Tics Scale (PUTS) | Part 1: days 0, 14, 28, 42, 56; Part 2: days 0, 14, 28
  The Premonitory Urge for Tics Scale (PUTS) is a patient self-assessment of the intensity of agreement of several statements describing the unpleasant qualities of premonitory feelings preceding tics. Each statement is being rated on a scale from 1 (not at all) to 4 (very much). The total score is being calculated by summing the single scores. The range of the total score is between 9, corresponding to a minimal intensity of premonitory urges for tics and 36, an extremely high intensity with probable severe impairment.
Clinical Global Impressions Scale for Improvement (CGII) | Part 1: days 14, 28, 42, 56; Part 2: days 14, 28
  The Clinical Global Impression of Improvement (CGI-I) is a 7-point ordinal, clinician-rated scale used to assess patients' overall improvement in disease status relative to their condition at baseline. A rating of 1 indicates a very much improved condition, compared to the subject's prior condition, while a rating of 7 means a very much worse condition respectively.
AE occurrence | Throughout the study: Part 1: day - 30 to day 70; Part 2: day 0 to day 42
  All Adverse Events (AE) occurring during the clinical trial will be registered, documented and evaluated.
SAE occurrence | Throughout the study: Part 1: day - 30 to day 70; Part 2: day 0 to day 42
  All Serious Adverse Events (SAE) occurring during the clinical trial will be registered, documented and evaluated.
SUSAR occurrence | Throughout the study: Part 1: day - 30 to day 70; Part 2: day 0 to day 42
  All Serious Unexpected Serious Adverse Reactions (SUSAR) occurring during the clinical trial will be registered, documented and evaluated.
Discontinuations due to AE occurrence | Throughout the study: Part 1: day - 30 to day 70; Part 2: day 0 to day 42
  All discontinuations due to (Adverse Events) AE occurring during the clinical trial will be evaluated.

CONTACTS AND LOCATIONS:
Overall Officials: Chan Beals, M.D., Ph.D., Study Director — Abide Therapeutics, Inc.
Locations (8):
- Germany (5):
  - Charité, Universitätsmedizin Berlin, Klinik für Neurologie mit Experimenteller Neurologie, Berlin
  - Uniklinik Köln, Klinik für Psychiatrie und Psychotherapie, Cologne
  - Medizinische Hochschule Hannover (MHH), Klinik für Psychiatrie, Sozialpsychiatrie und Psychotherapie, Hanover
  - Universität zu Lübeck, CBBM / Institut für Neurogenetik, Lübeck
  - LMU Klinikum der Universität München, Klinik für Psychiatrie und Psychotherapie, München
- Centrum Medyczne Damiana Holding Sp zo.o., Warsaw, Poland
- Spain (2):
  - Complejo Hospitalario Regional Virgen Del Rocío, Seville, Andalusia
  - Complejo Hospitalario Gregorio Marañón, Madrid

REFERENCES:
- [Derived] Muller-Vahl KR, Fremer C, Beals C, Ivkovic J, Loft H, Schindler C. Monoacylglycerol Lipase Inhibition in Tourette Syndrome: A 12-Week, Randomized, Controlled Study. Mov Disord. 2021 Oct;36(10):2413-2418. doi: 10.1002/mds.28681. Epub 2021 Jun 12. PMID 34117788